CLINICAL TRIAL: NCT02627170
Title: Measurements of Corneal Biomechanical Properties Using a Dynamic Scheimpflug Analyzer for Normal Adults in South Korea
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0943
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy adults group: Age 20 to 40 years of age and have myopia with a spherical equivalent (SE) between 0.00 and -11.00 diopters (D)
  Interventions: Device: dynamic Scheimpflug analyzer (corneal visualization Scheimpflug technology [Corvis ST], OCULUS, Wetzlar, Germany)

INTERVENTIONS:
Device: dynamic Scheimpflug analyzer (corneal visualization Scheimpflug technology [Corvis ST], OCULUS, Wetzlar, Germany)

SUMMARY:
The human cornea is affected by the magnitude and velocity of both internal and external forces because the cornea has both static and dynamic resistance components. Considering these natures of the human cornea, many investigators have tried to demonstrate corneal biomechanical properties to understand these characteristics of the cornea. Corneal biomechanical properties are known to influence the accuracy of measurements in intraocular pressure (IOP) and are recognized as important factor to explain the susceptibility of development of glaucomatous damage. Until recently, the only instrument which enabled the in vivo measurements of the ocular biomechanical properties was ocular response analyzer (ORA, Reichert Ophthalmic Instruments, Depew, NY, USA).8 The ORA has been used to assess the biomechanical properties of the cornea according to the dynamic bidirectional applanation process. A dynamic Scheimpflug analyzer (corneal visualization Scheimpflug technology [Corvis ST], OCULUS, Wetzlar, Germany) has been introduced recently and has become a useful instrument for evaluating corneal biomechanical properties. The dynamic Scheimpflug analyzer captures the dynamic process of corneal deformation caused by an air puff using an ultra-high-speed Scheimpflug camera at a rate of up to 4,330 images per second. Until now, well-organized analysis on the normative data of the corneal biomechanical profiles measured with the dynamic Scheimpflug analyzer has not been reported yet. Hence, in the present study, we aim to conduct normative data analysis for the corneal biomechanical properties with the dynamic Scheimpflug analyzer in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Only the participants age > 20 years old were included
* have myopia with a spherical equivalent (SE) between 0.00 and -11.00 diopters (D)

Exclusion Criteria:

* Participants were excluded from analyses if they had abnormal eye-related findings except for clinically insignificant senile cataract, previous ocular or intraocular surgery, glaucoma, history of ocular diseases such as glaucoma or age-related macular degeneration, presence of corneal abnormalities such as keratoconus and forme fruste keratoconus, or corneal scarring that would preclude accurate measurements.
* Participants with diabetes mellitus were also excluded, because of the possible effects of the disease on corneal hysteresis.None of the participants were using eye drops, especially anti-IOP agents, which can change the biomechanical properties of the cornea

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal healthy population
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
applanation time (AT) | 1 hour
applanation length (AL) | 1 hour
corneal velocity (CV) | 1 hour
deformation amplitude | 1 hour
peak distance | 1 hour
radius | 1 hour
maximal concave power | 1 hour
central corneal thickness (CCT) | 1 hour
intraocular pressure (IOP) | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
undecided yet